CLINICAL TRIAL: NCT02419586
Title: Effectiveness of Gum Chewing on Reduction of Postoperative Paralytic Ileus for Chinese Colorectal Cancer Patients Underwent Laparoscopic Colorectal Surgery and Enhanced Recovery Program
Brief Title: Effectiveness of Gum Chewing on Ileus in Chinese Colorectal Patients Underwent Laparoscopic Colorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shum Nga Fan (Other Government)
Responsible Party: Sponsor-Investigator, Shum Nga Fan, APN, Hospital Authority, Hong Kong
Organization: Hospital Authority, Hong Kong (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CRC03
Record Dates: First submitted 2015-03-04; First posted 2015-04-17 (Estimated); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- bubble gum chewing and routine care (Experimental): Start chewing gum on postoperative day at three times daily with no more than 30 minutes till discharged
  Interventions: Other: bubble gum
- routine care (No Intervention): Non interventional group will receive existing routine care as usual

INTERVENTIONS:
Other: bubble gum — Chewing gum group patients performing gum chewing on postoperative day 1 at three times daily for 30 minutes after operation and until discharged.
  Arms: bubble gum chewing and routine care

SUMMARY:
Gum chewing group will have less ileus and early resume of bowel motion than control group.

DETAILED DESCRIPTION:
The standardize surgical techniques, less used of epidural analgesia, early ambulation and used of naso-gastric tube for decompression are aimed to reduce the paralytic ileus after abdominal surgery . Most Western studies have examined and found that gum chewing are able to prevent postoperative ileus or promotes early bowel function after abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed colorectal cancer undergoing laparoscopic resection in in Queen Mary Hospital
* At least 18 years
* Speak Cantonese
* Able to follow study protocol and chewing gum study

Exclusion Criteria:

* Cognitive disability
* Requirement of epidural analgesia
* Requirement of intensive care unit/ High dependency unit care postoperatively
* Inability to chew
* Presence of procedure other than colorectal resection
* Non Chinese

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Time to first flatus | from postoperative day 0 till an expected average of day 7
  Time to passage of flatus after surgery was significantly shorter in the intervention group (22 vs 39 hours, p=0.007).

SECONDARY OUTCOMES:
Time to first sense of hunger | from postoperative day 0 till an expected average of day 7
  Patients in the intervention group also noticed feeling of hunger earlier (17 vs 40 hours, p<0.001).
Time to first bowel movement, | from postoperative day 0 till an expected average of day 7
  The first bowel motion also occurred earlier in the intervention group (22 vs 52 hours, p<0.001)
Length of stay | from postoperative day 0 till an expected average of day 7
  There is no difference in length of stay between intervention group or control group

CONTACTS AND LOCATIONS:
Overall Officials: Nga Fan Shum, Principal Investigator — Hospital Authority, Queen Mary Hospital
Locations (1):
- Queen Mary Hospital, Hong Kong, China

REFERENCES:
- [Derived] Shum NF, Choi HK, Mak JC, Foo DC, Li WC, Law WL. Randomized clinical trial of chewing gum after laparoscopic colorectal resection. Br J Surg. 2016 Oct;103(11):1447-52. doi: 10.1002/bjs.10277. PMID 27654648